CLINICAL TRIAL: NCT03990298
Title: Prospective Use of Awake Endoscopy to Direct Inspire Therapy for Obstructive Sleep Apnea
Brief Title: Prospective Use of Awake Endoscopy for Inspire Activation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 828956
Record Dates: First submitted 2019-05-23; First posted 2019-06-18 (Actual); Results first posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- All subjects (Other): Awake endoscopic exam will be performed to measure airway size in the retropalatal and retroglossal upper airway regions using different Inspire implant configurations and voltages.
  Interventions: Diagnostic Test: Awake endoscopy

INTERVENTIONS:
Diagnostic Test: Awake endoscopy — Awake endoscopic exam will be performed to measure airway size in the retropalatal and retroglossal upper airway regions using different Inspire implant configurations and voltages. The optimal test configuration determined on endoscopy will be tested during a sleep study and compared to the standard-of-care device configuration, with improvements in sleep study outcomes indicating that awake endoscopy is useful during Inspire implant activation.

SUMMARY:
The aim of this study is to examine a new method of device configuration for the Inspire upper airway stimulator. First, the investigators will attempt to determine optimal configuration by quantifying changes in upper airway size with different implant configurations using awake nasal endoscopy. The configuration/voltage that results in the greatest increase in upper airway size and is tolerated by the patient will be selected. Participants will then undergo a sleep study so that increased airway size may be correlated with changes in sleep study parameters including AHI and oxygen desaturation index (ODI). Airway size and sleep study parameters using the standard device configuration (+-+)/voltage will be compared to airway size and sleep study parameters using the test, or "optimal," configuration/voltage to determine the usefulness of awake endoscopy in activation of the Inspire device.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe OSA who have undergone Inspire UAS implantation by the principal investigator
* Must have symptoms of OSA prior to Inspire implantation
* AHI between 15 and 65, where central and mixed apnea is 25% or more, and the level of collapse is in the soft palate area BMI less than 32
* Age 18 or above

Exclusion Criteria:

* Significant central sleep apnea
* Presence of other sleep disorders
* History of neurologic or neuromuscular disease
* Historical or present substance abuse
* Bleeding disorders
* Autoimmune diseases that increase risk of nasal trauma such as Wegener's, Sarcoidosis, etc.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-06-09 (Actual); Study Completion 2020-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erica Thaler, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Awake Endoscopic Exam: Awake endoscopic exam will be performed to measure airway size in the retropalatal and retroglossal upper airway regions using different Inspire implant configurations and voltages.
  Awake endoscopy: Awake endoscopic exam will be performed to measure airway size in the retropalatal and retroglossal upper airway regions using different Inspire implant configurations and voltages. The optimal test configuration determined on endoscopy will be tested during a sleep study and compared to the standard-of-care device configuration, with improvements in sleep study outcomes indicating that awake endoscopy is useful during Inspire implant activation.
Period: Overall Study
Arm/Group | Awake Endoscopic Exam
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Awake Endoscopic Examination: Subjects who underwent upper airway stimulation (UAS) implantation were recruited for a prospective single-arm cohort study during UAS device activation. Functional thresholds were recorded for all settings. Awake nasopharyngoscopy was performed to examine the retropalatal (RP) and retroglossal (RG) regions at rest and during activation at five different electrode configurations at their functional thresholds. Electrode configurations included: +-+, ---, -o-, o-o, and -+-. Cross-sectional measurements were made by two blinded reviewers and reported as percent change in airway size.
Arm/Group | Awake Endoscopic Examination
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.1 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Distribution of Electrode Configurations Resulting in Greatest Retropalatal Expansion Among Cohort Subjects
Description: The hypoglossal nerve stimulator has a triode (three electrodes) that is wrapped around the nerve. Each electrode can be configured to either "Off," "Positive," or "Negative." For each electrode configuration we determined the percentage of patients with the greatest retropalatal cross-sectional area resulting from stimulation.
Time Frame: One month after surgical implantation of UAS
Measure: Count of Participants; unit: Participants
Arm/Group | Awake Endoscopic Exam
Number analyzed (Participants) | 16
Participants
  Positive, Negative, Positive (+-+) | 7
  Negative, Negative, Negative (---) | 3
  Off, Negative, Off (o-o) | 3
  Negative, Off, Negative (-o-) | 2
  Negative, Positive, Negative (-+-) | 1

ADVERSE EVENTS:
Time Frame: 31 months
Groups:
- Awake Endoscopic Examination: Awake endoscopic exam will be performed to measure airway size in the retropalatal and retroglossal upper airway regions using different Inspire implant configurations and voltages.
  Awake endoscopy: Awake endoscopic exam will be performed to measure airway size in the retropalatal and retroglossal upper airway regions using different Inspire implant configurations and voltages. The optimal test configuration determined on endoscopy will be tested during a sleep study and compared to the standard-of-care device configuration, with improvements in sleep study outcomes indicating that awake endoscopy is useful during Inspire implant activation.
Arm/Group | Awake Endoscopic Examination
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-22): https://cdn.clinicaltrials.gov/large-docs/98/NCT03990298/Prot_SAP_000.pdf